CLINICAL TRIAL: NCT06496165
Title: Comparison of the Effects of Remimazolam Besylate and Propofol Sedation on Hemodynamic for Coronary Artery Bypass Graft Patients：a Prospective, Single Blinded, Randomized Controlled Trial
Brief Title: Remimazolam Besylate and Propofol Sedation on Hemodynamic for Coronary Artery Bypass Graft Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REMAP
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam (Experimental)
  Interventions: Drug: Remimazolam
- propofol (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Intravenous pump injection. The loading dose will be 0.1mg/kg, the maintenance dose will be 0.1-0.5mg/kg/h, with the target RASS be -2-0
  Arms: remimazolam
Drug: Propofol — Intravenous pump injection. The loading dose will be 0.5mg/kg, the maintenance dose will be 1-4mg/kg/h, with the target RASS be -2-0
  Arms: propofol

SUMMARY:
In the immediate postoperative period following cardiac surgery, many patients require short-term sedation until cardiovascular and respiratory stability has been achieved and weaning from artificial ventilation can be started. For these patients, current guideline recommended propofol over benzodiazepine, mainly because of the short elimination half life of propofol. However, hypotension, a very common side effect of propofol, may impose restrictions on its use in some cardiac surgery patients. Remimazolam besylate is a novel, ultra-short-acting benzodiazepine that undergoes organ-independent metabolism by tissue esterases into an inactive metabolite. In other words, remimazolam has both the property of quick offset of effect like propofol and the stable hemodynamic effect like midazolam, making it favorable for use as a sedative in cardiac surgery patients. The aim of this study is to evaluate the hemodynamic effect of remimazolam besylate versus propofol in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form voluntarily and follow the plan requirements;
* age over 60 years old;
* post coronary artery bypass surgery;
* anticipated mechanical ventilation duration >8 hours
* admission to the cardiac surgery intensive care unit of Zhongshan hospital, Fudan University

Exclusion Criteria:

* delirium before surgery
* severe cognitive dysfunction before surgery
* patients with over degree II A-V block or consistent bradycardia
* patients who are still not awake 12 hours after surgery
* patients who are agitated or cannot follow command
* patients with mechanical circulatory support (ECMO, IABP)
* patients who are allergy to propofol or remimazolam
* BMI≥30kg/m2
* patients with much drainage, the surgery ask for blood pressure control or reopen the chest

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of hypotension during infusion of remimazolam or propofol in patients undergoing coronary artery bypass surgery | Within 8 hours of study drug used

SECONDARY OUTCOMES:
RASS score during infusion of remimazolam or propofol in patients undergoing coronary artery bypass surgery | Within 8 hours of study drug used

OTHER OUTCOMES:
rate of delirium during infusion of remimazolam or propofol in patients undergoing coronary artery bypass surgery | Within 8 hours of study drug used

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan university, Shanghai, Shanghai Municipality, China